CLINICAL TRIAL: NCT05440942
Title: A Phase 1 Trial of Combined MEK, STAT3 and PD-1 Inhibition in Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Combined MEK, STAT3 and PD-1 Inhibition in Metastatic Pancreatic Ductal Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peter Hosein, MD (Other)
Collaborators: Incyte Corporation (Industry); Novartis Pharmaceuticals (Industry); University of Miami Sylvester Comprehensive Cancer Center (Other)
Responsible Party: Sponsor-Investigator, Peter Hosein, MD, Associate Professor of Clinical, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20220171
Record Dates: First submitted 2022-06-27; First posted 2022-07-01 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — trametinib; ruxolitinib

STUDY DESIGN:
Intervention Model Description: Phase 1 dose escalation/de-escalation and dose expansion design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part 1 Schedule A: TR^2 Dose Escalation/De-Escalation (Experimental): Participants in this group will receive Trametinib, Ruxolitinib and Retifanlimab in a dose escalation/de-escalation design to determine the maximum tolerated dose (MTD). Participants will receive Trametinib and Ruxolitinib for two weeks on (Days 1-14) and two weeks off (Days 15-28) and Retifanlimab on Day 8 of a 28-day cycle. Doses will be administered as follows:
  * Dose Level -1A: Trametinib 1 mg orally (PO), Ruxolitinib 5 mg PO, Retifanlimab 500 mg intravenously (IV);
  * Starting Dose Level 1A: Trametinib 1.5 mg PO, Ruxolitinib 10 mg PO, Retifanlimab 500 mg IV;
  * Dose Level 2A: Trametinib 2 mg PO, Ruxolitinib 10 mg PO, Retifanlimab 500 mg IV;
  * Dose Level 3A: Trametinib 2 mg PO, Ruxolitinib 15 mg PO, Retifanlimab 500 mg IV.
  Interventions: Drug: Trametinib; Drug: Ruxolitinib; Drug: Retifanlimab
- Part 1 Schedule B: TR^2 Alternate Schedule (Experimental): Participants in this group will receive the MTD determined in Part 1 Schedule A on a continuous dosing cycle: Trametinib and Ruxolitinib on Days 1-28 and Retifanlimab on Day 8 of a 28-Day Cycle.
  Interventions: Drug: Trametinib; Drug: Ruxolitinib; Drug: Retifanlimab
- Part 2: TR^2 Expansion Cohort (Experimental): Participants in this group will receive Trametinib, Ruxolitinib and Retifanlimab at the most appropriate dose and schedule determined in Part 1. Participants will continue to receive treatment as long as receiving clinical benefit or until disease progression.
  Interventions: Drug: Trametinib; Drug: Ruxolitinib; Drug: Retifanlimab

INTERVENTIONS:
Drug: Trametinib — Trametinib will be administered orally once daily via tablet.
  Other Names: GSK1120212; TMT212-NXA; Mekinist
Drug: Ruxolitinib — Ruxolitinib will be administered orally twice daily (BID) via tablet.
  Other Names: INCB018424; INC424
Drug: Retifanlimab — Retifanlimab will be administered intravenously (IV) on Day 8 of a 28-day cycle..
  Other Names: INCMGA00012

SUMMARY:
The purpose of this research is to test whether a combination treatment of Trametinib, Retifanlimab, and Ruxolitinib (TR^2) will reduce tumor size in patients with metastatic pancreatic ductal adenocarcinoma (PDAC).

DETAILED DESCRIPTION:
Adenocarcinoma of the pancreas (PDAC) remains a major therapeutic challenge due to its innate and acquired chemoresistance. Three major contributors to therapeutic resistance that have been difficult to overcome in PDAC are mutations in the KRAS oncogene, the presence of a dense desmoplastic stroma that acts as a barrier to drug delivery and effector immune cell infiltration, and the immunosuppressive tumor microenvironment (TME) that renders the tumor innately resistant to immunotherapy.

The Merchant and Datta labs at the University of Miami (UM) has extensively studied the targeting of downstream effectors of oncogenic RAS. They have shown that mitogen-activated extracellular signal-regulated kinase inhibition (MEKi) results in reciprocal activation of signal transducer and activator of transcription 3 (STAT3) signaling, which confers therapeutic resistance and continued PDAC cell growth. Combined inhibition of Janus kinases (JAK)/STAT3 (STAT3i) and MEKi overcomes therapeutic resistance following RAS inhibition that is mediated through parallel feedback loop activation.

They have also identified a novel mechanism showing that combined MEKi and STAT3i also inhibits tumor fibrosis and enhances CD8+ cytotoxic T-cell (CTL) infiltration to the tumor while downregulating immunosuppressive regulatory T cells (Tregs) and myeloid derived suppressor cells (MDSCs) in the TME, resulting in reduced tumor burden and improved survival in genetically engineered mouse models of PDAC.

Furthermore, they have shown that the anti-tumor effects of MEKi and STAT3i are T-cell dependent. This change in the TME, however, is accompanied by sustained PD-L1/PD-1 and cytotoxic T lymphocyte antigen-4 (CTLA-4) expression. The preliminary results further demonstrate that combined MEKi and STAT3i with PD-1 inhibition can harness the effects of immune checkpoint inhibitors for an enhanced anti-tumor response.

Based on many years of preclinical investigation, this triplet combination appears to be a promising option and this clinical trial will tests its safety and effectiveness in patients with metastatic PDAC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, metastatic pancreatic adenocarcinoma. Patients with adenosquamous carcinoma and mixed adenocarcinoma/neuroendocrine carcinoma (MANEC) of the pancreas are eligible, but pure neuroendocrine neoplasms are excluded.
2. Progression of disease or intolerance to at least one standard line of chemotherapy.

   1. Patients who are candidate for an anti-PD-1 antibody due to Microsatellite instability -High (MSI-H) or tumor mutational burden (TMB)-high status must have been treated with this drug before being eligible for this trial.
   2. Prior treatment with an anti-PD(L)-1 antibody is allowed unless this therapy was stopped due to an immune-related adverse event.
   3. Patients who are candidate for a poly (ADP-ribose) polymerase (PARP) inhibitor due to a germline BRCA1/2 mutation must have been treated with this drug before being eligible for this trial.
3. At least one tumor measurable by CT scan. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or >10 mm with spiral CT scan.
4. Adult patients (≥ 18 years of age).
5. Male or non-pregnant and non-lactating female. Men and women with intact reproductive potential must agree to use contraception as outlined in Section 4.9.
6. Adequate biological parameters as demonstrated by the following blood counts at Screening (obtained ≤ 21 days prior to enrollment) and at Baseline-Day 0:

   1. Absolute neutrophil count (ANC) ≥ 1.0 × 10^9 cells/L.
   2. Platelet count ≥ 100,000 cells/mm3 (100 × 10^9 cells/L).
   3. Hemoglobin (Hgb) ≥ 9 g/dL.
7. Adequate blood chemistry levels at Screening (obtained ≤ 21 days prior to enrollment) and at Baseline-Day 0:

   1. Aspartate aminotransferase (AST) - serum glutamic-oxaloacetic transaminase (SGOT); alanine transaminase (ALT) - serum glutamic-pyruvic transaminase (SGPT) ≤ 2.5 × upper limit of normal (ULN) range, unless liver metastases are present, then ≤ 5 × ULN is allowed.
   2. Total bilirubin ≤ 1.5 × ULN.
   3. Estimated creatinine clearance of > 60 mL/min (per Cockcroft-Gault formula).
   4. Albumin ≥ 3.0 g/dL.
8. Eastern Cooperative Oncology Group (ECOG) performance status from 0 to ≤ 1 (see APPENDIX A: PERFORMANCE STATUS SCALES).
9. At least two weeks since the last anti-cancer therapy (e.g., chemotherapy, radiation therapy).
10. All toxicities from the last anti-cancer therapy should be resolved to < grade 1.
11. Patient has been informed about the nature of the study, has agreed to participate in the study, and signed the Informed Consent Form (ICF) prior to participation in any study-related activities.

Exclusion Criteria:

1. Patients with pure neuroendocrine neoplasms of the pancreas.
2. Brain metastases.
3. Uncontrolled ascites.
4. Increase of ECOG to > 1 between screening and enrollment.
5. Corrected QT interval (QTcF) > 450 msec.
6. Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
7. History of HIV and/or Hepatitis B or C infection.
8. History of active autoimmune disease that, in the opinion of the Investigator, could deteriorate upon treatment with an immune checkpoint inhibitor.
9. Concurrent use of systemic corticosteroids equivalent to or greater than prednisone 10 mg/day within two weeks of start of study therapy.
10. Receipt of a live vaccine within 30 days prior to enrollment.
11. Patients who are not up to date on FDA-approved coronavirus disease 2019 (COVID-19) vaccination series will be excluded.
12. Any impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or extensive small bowel resection).
13. History of interstitial lung disease or pneumonitis.
14. History of liver disease as follows:

    1. Cirrhosis
    2. Autoimmune hepatitis
    3. Portal hypertension
    4. Drug-induced liver steatosis
15. Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, including any of the following:

    1. History of myocardial infarction, angina pectoris, symptomatic pericarditis, or coronary artery bypass graft within six months prior to study entry
    2. Documented cardiomyopathy
    3. Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO)
16. Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome or any of the following risk factors for Torsades de Pointe, including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia.
17. Concomitant medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued or replaced by safe alternative medication (e.g., within five half-lives or seven days prior to starting study drug).
18. Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade arterioventricular block (e.g., bifascicular block, Mobitz type II, and third-degree atrioventricular block).
19. Treatment refractory hypertension defined as a blood pressure of systolic blood pressure (SBP) >140 mmHg and/or diastolic blood pressure (DBP) > 90 mm Hg that cannot be controlled by anti-hypertensive therapy.
20. A history or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR) including:

    1. Presence of predisposing factors to RVO or CSR (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled hypertension, uncontrolled diabetes mellitus, or a history of hyperviscosity or hypercoagulability syndromes); or
    2. Visible retinal pathology as assessed by ophthalmic examination that is considered a risk factor for RVO or CSR.
21. Currently receiving any of the following substances and cannot be discontinued seven days prior to Cycle 1 Day 1:

    1. Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pomelos, star-fruit, and Seville oranges.
    2. Substances that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5.
    3. Herbal preparations/medications and/or dietary supplements.
22. History of allergy or hypersensitivity to any of the study drugs, their pharmaceutical class, or any of their excipients.
23. Concomitant serious medical or psychiatric illness that, in the opinion of the investigator, could compromise the patient's safety or integrity of the study data.
24. Concurrently enrolled in any other interventional clinical protocol or investigational trial involving administration of antineoplastic compounds for the treatment of metastatic pancreatic cancer.
25. Patient is unwilling or unable to comply with study procedures.
26. Patients with impaired decision-making capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | Up to 6 months
  The RP2D of combination therapy of trametinib, ruxolitinib and retifanlimab (TR^2) therapy will be determined as the maximum tolerated dose of combination treatment (in mg) as assessed by treating physician using the NCI-CTCAE Version 5.0.

SECONDARY OUTCOMES:
Incidence of Treatment-Related Toxicity | Up to 2 years
  The incidence of treatment-related dose limiting toxicities (DLTs), serious adverse events (SAEs) and Grade 3 or higher adverse events (AEs) in study participants receiving combination TR^2 therapy will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, per physician discretion.
Overall Survival (OS) | Up to 3 years
  Overall survival (OS) is defined as the elapsed time from study treatment initiation to death or date of censoring. Participants alive or those lost to follow-up will be censored at the last date known to be alive. OS rate will be reported as the percentage of participants still alive after start of treatment.
Percentage of Participants Achieving Overall Response | Up to 2 years
  Overall response will be determined as the percentage of participants achieving complete response (CR) or partial response to combination TR^2 treatment. Response will be assessed by treating physician using the revised Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hosein, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Laboratory evidence that led to the development of this clinical trial (currently under peer review) — https://www.biorxiv.org/content/10.1101/2021.03.07.434236v2